CLINICAL TRIAL: NCT03359434
Title: Impact of Blood Pressure Measurement Methods for the Prediction of Intracranial Hemorrhage After Thrombectomy in Acute Stroke
Brief Title: Blood Pressure Measurement Methods and Prediction of Intracranial Hemorrhage After Thrombectomy in Stroke
Acronym: BP-METROLOGY
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMI_2017_12
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Acute Stroke; Blood Pressure; Cerebral Hemorrhage
Keywords: Acute Stroke; Blood Pressure; Cerebral Hemorrhage
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Two measuring methods of blood pressure
  Interventions: Device: Clearsight device (Edwards) around the finger; Device: Intermittent blood pressure measurements with cuff.

INTERVENTIONS:
Device: Clearsight device (Edwards) around the finger — Continuous measurement of blood pressure with the Clearsight device (Edwards) around the finger, within 24 hours after reperfusion:
Device: Intermittent blood pressure measurements with cuff. — Standard method: 35 blood pressure measurements with cuff within 24 hours after reperfusion

SUMMARY:
A monocentric, non-randomized, prospective study in which each patient is his/her own control.

The study investigates 2 methods of blood pressure measurement, within the first 24 hours after reperfusion, i) Continuous measurement of blood pressure with the Clearsight device (Edwards) and ii) intermittent blood pressure measurements with cuff.

DETAILED DESCRIPTION:
Patients will be followed for 72 hours:

* inclusion after reperfusion: clinical evaluation with NIHSS (National Institute of Health Stroke Score) score, measurement of blood pressure.
* within 24 hours after reperfusion: blood pressure measurements
* at 24 hours: NIHSS score.
* Between 24 and 36 hours :cerebral scan (assessment of hemorrhagic transformations and cerebral infarction volumes).
* 72 hours after reperfusion: brain scanner in case of hyperdensity on the initial scanner

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Treated for occlusion of the internal carotid arteries and/or proximal middle cerebral arteries (M1 and M2 segments), vertebral artery, and/or basilar artery
* Affiliated with or beneficiary of a Social Security plan
* Having received informed information about the study and having given consent to participate in the study

Exclusion Criteria:

* Per-procedure hemorrhagic complications (before reperfusion is achieved)
* Patient benefiting from legal protection measures
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thrombectomy after acute stroke
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Occurence of intracranial hemorrhagic complications | 36 hours after baseline
  number of intracranial hemorrhagic complications (symptomatic or asymptomatic) on brain scanner, evaluated with a double centralized blind reading

CONTACTS AND LOCATIONS:
Overall Officials: MAZIGHI Mikael, MD PhD, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation Ophtalmologique A de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided